CLINICAL TRIAL: NCT06149546
Title: Exploring the Impact of a Multi-modal Nutritional Intervention in Patients Undergoing Chemotherapy for Pancreatic Cancer (FEED Trial)
Acronym: FEED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CTRIAL-IE 20-26
Record Dates: First submitted 2023-10-11; First posted 2023-11-29 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer; Multi-modal Nutritional
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Experimental): * High protein, high energy diet
  * Fish oil supplement (ProSure®)
  * Pancreatic Enzymes (Creon®)
  * A daily individualised step target (10% above your own baseline)
  * Four scheduled appointments with a dietitian
  Interventions: Dietary Supplement: Control
- Intervention (Experimental): * High protein, high energy diet
  * Fish oil supplement (ProSure®)
  * Pancreatic Enzymes (Creon®)
  * A daily individualised step target (10% above your own baseline)
  * Seven scheduled appointments with a dietitian
  * Six scheduled appointments with a physiotherapist
  Interventions: Dietary Supplement: Intervention

INTERVENTIONS:
Dietary Supplement: Control — * High protein, high energy diet
  * Fish oil supplement (ProSure®)
  * Pancreatic Enzymes (Creon®)
  * A daily individualised step target (10% above your own baseline)
  * Four scheduled appointments with a dietitian
  Arms: Control
Dietary Supplement: Intervention — * High protein, high energy diet
  * Fish oil supplement (ProSure®)
  * Pancreatic Enzymes (Creon®)
  * A daily individualised step target (10% above your own baseline)
  * Seven scheduled appointments with a dietitian
  * Six scheduled appointments with a physiotherapist
  Arms: Intervention

SUMMARY:
The study will examine if a multi-modal nutritional care package, with or without resistance training delivered with neoadjuvant chemotherapy, is effective at preventing loss of muscle strength during neoadjuvant chemotherapy for pancreatic cancer. There are two arms in this study: Control Arm will receive standard dietetic care and be prescribed standard pancreatic enzyme replacement therapy and oral nutritional supplement drinks with their neoadjuvant chemotherapy. The intervention Arm will have 3 additional dietitian visits and 6 physiotherapist visits that the control group will not.

DETAILED DESCRIPTION:
This is a translational, single-site, open-label, randomised, prospective 12-week study. 70 (35 in each arm) patients will be enrolled in the study; The study will examine if a multi-modal nutritional care package, with or without resistance training delivered concurrently to neoadjuvant chemotherapy, is effective at preventing loss of muscle strength during neoadjuvant chemotherapy for pancreatic cancer. There are two arms in this study: The control group will receive standard dietetic care and be prescribed standard pancreatic enzyme replacement therapy and oral nutritional supplement drinks concurrently with their neoadjuvant chemotherapy. The intervention group in comparison to the control group will have 3 additional dietitian visits and 6 physiotherapist visits that the control group will not.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give signed informed consent and willing and able to comply with the protocol.
2. Patients aged 18 years and above.
3. Patients with newly diagnosed, pathologically confirmed pancreatic ductal adenocarcinoma who will undergo neoadjuvant chemotherapy following formal MDT assessment at St Vincent's University Hospital, specifically FOLFIRINOX or Gemcitabine with Nab-Paclitaxel (and/or any additional therapy regimen approved by NCCP).
4. Patients have CT scan available and suitable for body composition analysis within 8 weeks prior to randomisation.
5. Patients have adequate upper limb dexterity to allow assessment of hand grip strength.

Exclusion Criteria:

1. Patients who are unable to consume oral diet and require prolonged enteral and/or parenteral nutritional support.
2. Patient with any significant history of non-compliance to medical treatments or with inability to grant reliable informed consent.
3. Patients who can/will not consume fish and pork products due to allergy, intolerance, religious beliefs, or dietary preferences.
4. Patients with known blood clotting disorders, e.g antiphospholipid syndrome, factor V Leiden syndrome, haemophilia /any liver disease which has progressed to liver cirrhosis where prolonged fish oil supplementation is unsafe.
5. Patients with uncontrolled hypertension (BP >180/110 mm Hg) which prohibits exercise.
6. Patients with muscle wasting disorders, e.g. paraplegia, motor neuron disease, Duchenne muscular dystrophy, multiple sclerosis.
7. Women who are pregnant or breastfeeding due to differing nutritional needs and macronutrient metabolism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of a multi-modal nutrition-led intervention in preventing loss of muscle strength (hand-grip strength) during chemotherapy | 12 weeks
  To compare the effectiveness of a multi-modal nutrition-led intervention in preventing loss of muscle strength (Percentage change in handgrip strength as determined by handgrip dynamometry) during chemotherapy with an intensive multi-modal nutrition and physiotherapist delivered intervention (1:1 randomisation).

SECONDARY OUTCOMES:
Effectiveness of the intervention compared to the control on weight changes | 12 weeks
  To compare the effectiveness of a multi-modal nutrition-led intervention on weight changes (kg and %) versus the control.
To compare the effectiveness of the intervention compared to the control on treatment delivery | 6 months
  Treatment delivery will be defined based on the occurrence of dose limiting toxicity (NCI CTCAE grading V5).
To compare the effectiveness of the intervention compared to the control on treatment delivery | 6 months
  Treatment delivery will be defined based on the need for dose reduction due to weight loss.
To compare the effectiveness of the intervention compared to the control on treatment delivery | 6 months
  Treatment delivery will be defined based on unplanned hospital admissions (frequency, duration (days), reason).
To compare the effectiveness of the intervention compared to the control on treatment response | 6 months
  Treatment response will be assessed by Resectability Status per National Cancer Control Network (NCCN)
To compare the effectiveness of the intervention compared to the control on treatment response | 6 months
  Treatment response will be assessed by Radiographic Classification of Borderline Resectable Pancreatic Cancer
To compare the effectiveness of the intervention compared to the control on patient acceptance/adherence. | 12 weeks
  Patient acceptance/adherence is defined as attendance at dietetic and physiotherapy appointments, dose of ONS and PERT delivered vs prescribed, step target achievement, exercise program adherence and progress.
Patient health-related quality of life (change in EORTC QLQ-C30 function or symptom score) | 12 weeks
  To compare the effectiveness of a multi-modal nutrition-led intervention on patient health-related quality of life (change in European Organisation for Research and Treatment of Cancer - Core Quality of Life questionnaire (EORTC QLQ-C30) function or symptom score) versus the control.
  The core EORTC QLQ C30 questionnaire has five functioning subscale scores and nine symptoms subscale scores.
  Minimum value = 0; Max value = 100 Function Scales: Higher numbers mean better function Symptom Scale: Higher numbers mean more symptoms
Change in Timed-up and Go (seconds) between control and intervention cohorts. | 12 weeks
  To compare the effectiveness of a multi-modal nutrition-led intervention on function (change in Timed-up and Go (seconds)) versus the control.
Changes in inflammatory markers and cytokine levels between control and intervention cohorts. | 12 weeks
  Changes in C-reactive Protein (CRP) will be measured between control and intervention cohorts.
Changes in inflammatory markers and cytokine levels between control and intervention cohorts. | 12 weeks
  Changes in Tumour Necrosis Factor-alpha (TNF-α) will be measured between control and intervention cohorts.
Changes in inflammatory markers and cytokine levels between control and intervention cohorts. | 12 weeks
  Changes in Interleukin-6 (IL-6) will be measured between control and intervention cohorts.
Changes in lumbar skeletal muscle index between control and intervention cohorts. | 6 months
  To compare the effectiveness of a multi-modal nutrition-led intervention on lumbar skeletal muscle index (cm²/m²) via diagnostic and restaging CT scans.
Changes in skeletal muscle between control and intervention cohorts. | 6 months
  To compare the effectiveness of a multi-modal nutrition-led intervention on skeletal muscle (area in cm²) via diagnostic and restaging CT scans
Changes in skeletal muscle between control and intervention cohorts. | 6 months
  To compare the effectiveness of a multi-modal nutrition-led intervention on skeletal muscle (mass in kg) via diagnostic and restaging CT scans
Effectiveness of the intervention compared to the control on body composition indices | 6 months
  To compare the effectiveness of a multi-modal nutrition-led intervention on lumbar adipose tissue (area in cm²) via diagnostic and restaging CT scans.
Effectiveness of the intervention compared to the control on body composition indices | 6 months
  To compare the effectiveness of a multi-modal nutrition-led intervention on lumbar adipose tissue (mass in kg) via diagnostic and restaging CT scans.
Effectiveness of the intervention compared to the control on body composition indices | 6 months
  To compare the effectiveness of a multi-modal nutrition-led intervention on body composition indices: assessment of muscle attenuation (Hounsfield Units (HU)) via diagnostic and restaging CT scans.
Effectiveness of the intervention compared to the control on Overall Survival | 6 months
  Overall survival rate at 6 months following the first day of chemotherapy and median overall survival time.

CONTACTS AND LOCATIONS:
Overall Officials: Oonagh Griffin, Dr, Principal Investigator — SVUH/University College Dublin; Ray McDermott, Prof, Principal Investigator — St Vincent's University Hospital, Ireland
Locations (1):
- St Vincent's University Hospital, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Pseudo-anonymised data will be shared with research partner University College of Dublin for performance of the study.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Study duration
Access Criteria: IPD data will be shared for all patients who provide informed consent to participation in the study